CLINICAL TRIAL: NCT02413112
Title: Minimum Resistance Training Frequency: Effect on Motivation and Adherence to Train, Overall Health Status and Neuromuscular Performance
Brief Title: Get in Shape in the Team Research: Porukalla Kuntoon Tutkimus
Acronym: PoKu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Responsible Party: Principal Investigator, Simon Walker, Post-doctoral researcher, University of Jyvaskyla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OKM/70/626/2014
Record Dates: First submitted 2015-02-19; First posted 2015-04-09 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Aging; Muscle Strength
Keywords: Aging; Sarcopenia; Resistance training; Strength; Muscle mass
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Training once per week (Experimental): Subjects train once per week in the University gym. All training sessions are supervised by the researchers.
  Interventions: Behavioral: Resistance training
- Training twice per week (Experimental): Subjects train twice per week in the University gym. All training sessions are supervised by the researchers.
  Interventions: Behavioral: Resistance training
- Thrice per week (Experimental): Subjects train three times per week in the University gym. All training sessions are supervised by the researchers.
  Interventions: Behavioral: Resistance training
- Non-training Control group (No Intervention): Subjects continue with their normal daily lives, just performing measurements

INTERVENTIONS:
Behavioral: Resistance training — Whole-body resistance training in the University gym that is supervised by researchers.
  Training once per week, Training twice per week, Training thrice per week.
  Arms: Thrice per week; Training once per week; Training twice per week

SUMMARY:
It is well accepted that physical activity in the form of resistance training produces a wide variety of neuromuscular-skeletal and health benefits. It is recommended in Finland that older individuals (over 65yr) should perform resistance training twice per week.

Unfortunately, only approx. 5% of older individuals fulfill this recommendation. As Finnish society grows ever older, research should focus on the specific needs of this group and how to improve participation in physical activity, which may ultimately lead to modification of physical activity recommendations - resistance training recommendations are currently the same for young and older adults and do not include specific recommendations on the type of resistance training. However, these recommendations appear to have been developed for "best possible" improvements in maximum strength and muscle size.

Therefore, it is of great importance to identify the number of resistance training sessions per week required to induce improvements in physical fitness, metabolic and bone health status, and importantly the reasons for adherence to/drop-out of resistance training interventions (e.g. motivation to train) in a multi-discipline study. This knowledge would benefit policy makers to update current recommendations for resistance training and to devise strategies to advise realistic targets for resistance training in the older, particularly the less-educated, age group (e.g. TELI-strategy for 2020).

The present study will include a 12-month resistance training intervention with a 12-month follow-up period. Interviews and questionnaires will assess psychological/sociological data and will be collected from both drop-out subjects and those that complete the intervention. Neuromuscular performance and functional capacity will be tested using conventional methods, along with body composition, bone density, and blood tests for metabolic markers of health. Diet and other physical activity will be controlled throughout the intervention period. Measurements are to be performed every 3 months.

It is expected that 5 international peer-reviewed articles will be published in 2016-2017. The data will be presented at international and national conferences in 2015-2017. Finally, results of the entire research will be published in national peer-reviewed journals (e.g. The Age Institute's "Raportteja"). All subjects will be invited to attend an information meeting where group results will be presented and explained.

ELIGIBILITY:
Inclusion Criteria:

* BMI<37
* Does not smoke
* Able to perform all tests and exercises
* Free from episodes during physical activity

Exclusion Criteria:

* BMI>37
* Use of waling aids
* Previous testosterone-altering treatment, e.g. in cancer treatment or hypogonadism
* Serious cardiovascular disease that may lead to complications during exercise
* Use of pharmaceuticals that affect neuromuscular or endocrine systems
* Regular endurance training>3hr per week
* Resistance training experience

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Force production (Isometric and dynamic maximum strength tests of lower limbs) | Change from baseline at 3, 9 and 15 months with data presented at 24 months post-initiation
  Isometric and dynamic maximum strength tests of lower limbs
Muscle hypertrophy (Cross-sectional area of quadriceps and triceps surae muscles) | Change from baseline at 3, 9 and 15 months with data presented at 24 months post-initiation
  Cross-sectional area of quadriceps and triceps surae muscles

SECONDARY OUTCOMES:
Body composition (DXA scanning) | Change from baseline at 3, 9 and 15 months with data presented at 24 months post-initiation
  for body fat and fat-free mass
Blood count | Change from baseline at 3, 9 and 15 months with data presented at 24 months post-initiation
  Basic blood count
Oral glucose tolerance test | Change from baseline at 3, 9 and 15 months with data presented at 24 months post-initiation
  Oral glucose tolerance test assessed for glucose and insulin concentrations
Basal hormone concentrations | Change from baseline at 3, 9 and 15 months with data presented at 24 months post-initiation
  Basal hormone concentrations from serum

CONTACTS AND LOCATIONS:
Overall Officials: Simon Walker, Ph.D, Principal Investigator — Univeristy of Jyvasklya